CLINICAL TRIAL: NCT06652789
Title: A Study to Evaluate the Efficacy of a Sleep Hygiene Behavior Intervention in Elderly With Insomnia
Brief Title: Efficacy of Sleep Hygiene Intervention in Elderly With Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Vishwajit Nimgaonkar, MD PhD, Pofessor of psychiatry and Human Genetics, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY23120054; 5D43TW009114-10 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Eelderly With Sleep Disturbances
Keywords: Sleep hygiene; Elderly; sleep disturbances
MeSH Terms: conditions — Sleep Hygiene; Parasomnias

STUDY DESIGN:
Intervention Model Description: Proposed study design: Interventional study (Pre-post study design) Elderly Out-patient and in-patients of Psychiatry department, St. John's Medical College and Hospital, Bengaluru, and St. John's Community Health Centre, Mugalur
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep hygiene teaching (Experimental): The intervention will be conducted over 6 weeks, and consist of engaging patients (and caregivers) in two 60-minute face to face sessions 3 weeks apart, and twice weekly telephonic follow ups lasting for 20 minutes each during the 6-week period.
  The 2 Direct face to face sessions will focus on health education about sleep. Each session will be conducted by a facilitator who has received training on the program, and will be delivered in a language that the participant is most fluent in (English/ Kannada/ Hindi/ Tamil/ Telugu). In case the participant is unable to come to the hospital for the session, the facilitator will visit the home of the patient to conduct the session (After taking consent)
  Interventions: Behavioral: Sleep hygiene

INTERVENTIONS:
Behavioral: Sleep hygiene — The intervention will be conducted over 6 weeks, and consist of engaging patients (and caregivers) in two 60-minute face to face sessions 3 weeks apart, and twice weekly telephonic follow ups lasting for 20 minutes each during the 6-week period.
  The 2 Direct face to face sessions in local language will focus on health education about sleep. (After taking consent)
  1. st session (60 mins) Information will be given about lifestyles that can affect sleep positively or negatively- adequate sleep time required for health, healthy and unhealthy sleep habits
  2. nd session Participants will be asked to indicate how many of the sleep hygiene techniques they were able to successfully implement since the previous session Successes and barriers will be discussed. provide solutions for standard difficulties faced Twice a week telephone calls. The participants will be followed up through telephonic conversation twice weekly with a gap of three to four days in between each call.

SUMMARY:
Sleep disorders are common among elderly, especially among those with mental health disorders. Impaired quality of sleep, in elderly, can lead to worsening of mental and physical health too. Due to high patient to doctor ratio in India and paucity of time in busy outpatients, there is inadequate information on causes of poor sleep quality in patients and a tendency to treat poor sleep with drugs. Studies on effectiveness of sleep hygiene techniques in insomnia also tend to exclude elderly. Thus, investigators have inadequate evidence on the applicability of such interventions in the elderly. In this study it is proposed to find the efficacy of a sleep hygiene behavioural intervention on severity of insomnia in elderly with sleep disturbances.

DETAILED DESCRIPTION:
Globally, the older population is increasing rapidly, and between 2015 and 2050, it is expected that the proportion of the world's population over 60 years will nearly double, from 12% to 22% (World Health Organization 2022).Untreated insomnia and other sleep disorders can have major health consequences (e.g., cardiovascular and metabolic disease, impaired cognitive functioning, and increased risk of psychiatric disorders, as well as an increased risk of accidents Studies have also shown that poor sleep is associated with increased risk of falls in the elderly Poor sleep quality has been shown to be associated with decline in cognitive function, impaired quality of life (QOL), excessive daytime sleepiness, fatigue, depression, increased mortality, economic burden, and possibly early institutionalization.

Insomnia is defined as "difficulty initiating sleep, difficulty maintaining sleep, morning awakening, or sleep that is chronically non-restorative or poor in quality, associated with daytime impairment such as fatigue, memory impairment, social or vocational dysfunction, or mood disturbance." There are several objective and subjective assessment tools for measuring sleep disorders, among which polysomnography (PSG) is the gold standard. Considering the time-consuming nature of PSG, associated expense and poor availability of it to most clinicians, it is generally not routinely used in the assessment of insomnia.

Studies have shown that people with insomnia engage in specific poor sleep hygiene practices, which may perpetuate insomnia. However, studies examining the effect of sleep hygiene practices on insomnia, illness severity and cognition are lacking in elderly patients. Sleep hygiene techniques can serve as a relatively inexpensive lifestyle intervention in elderly patients with insomnia. Sleep hygiene recommendations may be delivered using a variety of media and measures (print based, in person discussions, telephonic conversations, etc), resulting in increased access. In addition to being commonly used and readily available, sleep hygiene education does not necessarily require the direct involvement of a clinician and therefore can be widely disseminated, even to elderly persons or their caregivers, who may not seek medical treatment for their sleep problems.

Estimated required sample size:

n1 = 43 n2 = 43 n1 + n2 = 86

Formula used:

Where, σ - Pooled standard deviation d - Difference between 2 group means Z1-β - Z value for corresponding power Z1-α/2 - Two-sided Z value for corresponding α (1.96)

Description of Intervention The intervention will be conducted over 6 weeks, and consist of engaging patients (and caregivers) in two 60-minute face to face sessions 3 weeks apart, and twice weekly telephonic follow ups lasting for 20 minutes each during the 6-week period.

The 2 Direct face to face sessions will focus on health education about sleep. Each session will be conducted by a facilitator who has received training on the program, and will be delivered in a language that the participant is most fluent in (English/ Kannada/ Hindi/ Tamil/ Telugu). In case the participant is unable to come to the hospital for the session, the facilitator will visit the home of the patient to conduct the session (After taking consent).

1. st face to face session (60 mins) Participants (and caregivers if available) will be informed about the study once again.

   Information will be given about lifestyles that can affect sleep positively or negatively- adequate sleep time required for health, healthy and unhealthy sleep habits Proper nutrition and fluid intake, exercise, smoking, alcohol habits and their relation to sleep will be discussed Common sleep myths will be covered briefly The consequences of poor sleep will be explained The sleep hygiene intervention will have 14 simple steps to be followed by participants- 1) Food/snacks have to be consumed at least 2 hours before bed time 2) Avoid electronic gadget usage i.e., mobile phone, laptop for at least 1 hour before bedtime 3) Go to bed only when feeling sleepy and not before 4) Using the bedroom only for sleep or sexual activity 5) Getting out of bed if unable to fall asleep 6) Avoid fluid intake 1 hour before bedtime 7) Avoid caffeine 4 hours before bedtime 8) Avoid Alcohol/Smoking 2 hours before bedtime 9) Lights should be turned off/to very dim immediately after going to bed 10) Avoid planning for next day or future activities on bed 11) Do not look at the time if the sleep is disturbed in between 12) Maintain regular sleep and wake up time with maximum of ½ hour deviation 13) Avoid noisy environment after going to bed (avoid discussion/arguments/ loud songs) 14) Avoid fasting Participants will be asked to rate their confidence level of following the above steps on a scale from 1 (not at all confident) to 10 (completely confident). If the participant's rating is below 7, they will be asked to discuss perceived barriers to following the steps, ways to overcome them and increase their confidence level to a rating of at least 7.

   Participants will be provided with a booklet containing all of the information covered in the first session.
2. nd face to face session The session will start with participants being asked to summarize what they have learnt from the previous face to face session as well as weekly telephone calls Participants will be asked to indicate how many of the sleep hygiene techniques they were able to successfully implement since the previous session Successes and barriers faced during the previous month will be discussed. Facilitator will attempt to provide solutions for standard difficulties faced Participants will be reminded that not all recommendations may work for them. They will be encouraged to view the 6week period as an opportunity to discover approaches that will work for them personally.

Sleep hygiene techniques will be reiterated once again The session will also involve setting goals for the following 3 weeks based on performance during the previous month Twice a week telephone calls The participants will be followed up through telephonic conversation twice weekly with a gap of three to four days in between each call. Total 10 calls over 6-week period (only 1 call in the weeks where the face-to-face sessions are conducted, and this call will cover the points mentioned next under first call per week) Data Collection Tools A questionnaire including demographic characteristics and 6 standardized tools for assessment of sleep quality, depression, anxiety, cognitive status, quality of life, loneliness and pain severity will be used to collect the data for the study.

1. Socio-demographic data sheet in elderly: Will include name, age, sex, address, religion, education, occupation, income, marital status, presence of any co-morbidities, presence of any substance use, diagnosed psychiatric illness, duration of illness, medications the patient is on, participant's co-morbidities, list of medications that the participant is on, average number of time participant wakes up to pass urine (developed by the researchers).
2. Pittsburgh Sleep Quality Index (PSQI): The PSQI is a 19-item, self-rated questionnaire. It was developed by Buysse et al. to measure sleep quality and disturbance over the past month. It is intended to be used as a standardized sleep questionnaire in clinical settings. The 19 items are grouped into 7 components. Each of the sleep components is scored from 0 to 3, with 3 indicating the most dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
3. The Montreal Cognitive Assessment (MoCA): The MoCA was designed as a rapid screening instrument for assessment of cognitive impairment. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
4. Patient Health Questionnaire 9 (PHQ-9): The PHQ-9 is the nine-item depression scale of the patient health questionnaire. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. The PHQ-9 can function as a screening tool, an aid in diagnosis, and as a symptom tracking tool that can help track a patient's overall depression severity as well as track the improvement of specific symptoms with treatment.
5. Generalized Anxiety Disorder scale (GAD 7): The GAD-7 represents an anxiety measure based on seven items which are scored from zero to three. The whole scale score can range from 0 to 21 and cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
6. Short form of the revised UCLA Loneliness Scale: The scale consists of 3 items with response options hardly ever or never, some of the time and often. Responses to the items are summed to obtain the total scale score which ranges from 3 to 9 with higher scores indicating greater levels of loneliness (α = 0.72)
7. WHO Quality of Life Brief Questionnaire (WHOQoL BREF): It consists of 24 items to assess perception of quality of life in four domains, including physical health, psychological, social relationships and environment, and two items on overall QOL and general health. A higher score indicated a better QOL.
8. Visual Analogue Scale for Pain: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients
* Age 60 years and above
* With self-reported sleep disturbances, scoring >5 on PSQI
* Who speak and understand one of English/ Kannada/ Hindi/ Tamil/ Telugu

Exclusion Criteria:

* With delirium
* With terminal medical illness
* Parkinsons disease, dementia
* Patients with severe mental illness
* Clinically diagnosed obstructive sleep apnea
* Patients who fulfil ICD-10 criteria for Alcohol Dependence syndrome
* Patients who are on medications that interfere with sleep like hypnotics, anxiolytics, stimulants
* Patients who are on anti-depressants and antipsychotics
* Patients with restless leg syndrome.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Statistically significant change in PSQI score | Baseline and after one month
  Pre-and -post assessment by Pittsburgh Sleep Quality Index (PSQI).. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.

SECONDARY OUTCOMES:
Statistically significant change in PSQI score (Sustainability) | Baseline and after three month
  Pre-and -post assessment by Pittsburgh Sleep Quality Index (PSQI).. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Changes of pertinent measures | Baseline and after one month
  measures on the actigraphy device at 1 month movement over time to assess sleep and wakefulness
Changes of pertinent measures (sustainability) | Baseline and after three months
  measures on the actigraphy device at 3 months movement over time to assess sleep and wakefulness
Statistically significant change in cognitive impairment measured by The Montreal Cognitive Assessment (MoCA ) | Baseline and after one months
  The Montreal Cognitive Assessment (MoCA ) measures will be applied to measure cognive impairment. The Montreal Cognitive Assessment (MoCA) is a screening tool for mild cognitive impairment that's scored on a scale of 0 to 30 points. The total score is calculated by adding up the points from each task. A higher score indicates better cognitive function.
Statistically significant change cognitive impairment (sustainability) | Baseline and after three months
  The Montreal Cognitive Assessment (MoCA ) measures will be applied to measure cognive impairment. The Montreal Cognitive Assessment (MoCA) is a screening tool for mild cognitive impairment that's scored on a scale of 0 to 30 points. The total score is calculated by adding up the points from each task. A higher score indicates better cognitive function.
Statistically significant change in quality of life (WHO-QoL BREF score) | Baseline and after one month
  WHO Quality of Life Brief Questionnaire (WHOQoL BREF): It consists of 24 items to assess perception of quality of life . A higher score indicated a better QOL.
Statistically significant change in quality of life (WHO-QoL BREF score) (Sustainability) | Baseline and after three month
  WHO Quality of Life Brief Questionnaire (WHOQoL BREF): It consists of 24 items to assess perception of quality of life . A higher score indicated a better QOL.
Statistically significant change in pain | Baseline and after one month
  Visual Analogue Scale for Pain: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Statistically significant change in pain (sustainability) | Baseline and after three month
  Visual Analogue Scale for Pain: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Statistically significant change in Loneliness | Baseline and after one month
  Short form of the revised UCLA Loneliness Scale: The scale consists of 3 items with response options hardly ever or never, some of the time and often. Responses to the items are summed to obtain the total scale score which ranges from 3 to 9 with higher scores indicating greater levels of loneliness
Statistically significant change in Loneliness (Sustainability) | Baseline and after three month
  Short form of the revised UCLA Loneliness Scale: The scale consists of 3 items with response options hardly ever or never, some of the time and often. Responses to the items are summed to obtain the total scale score which ranges from 3 to 9 with higher scores indicating greater levels of loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Vishwajit L Nimgaonkar, MD, PhD, Principal Investigator — University of Pittburgh
Locations (1):
- St.John's Medical College and Hospital, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the trial as well as protocol will be shared on request at 1 years after results are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after publication of the study
Access Criteria: The study should be ethically approved and scientifically sound.